CLINICAL TRIAL: NCT05205447
Title: A Phase 1, Two-part, Open-label, Fixed-sequence Study to Evaluate the Effects of Multiple Doses of Itraconazole and Carbamazepine on the Single-dose Pharmacokinetics of LY3410738 in Healthy Adult Subjects
Brief Title: Study of the Effects of Itraconazole and Carbamazepine on LY3410738 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Data from part 2 no longer deemed necessary for this program.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-IDH-21005; I9Y-OX-JDHF (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-01-05; First posted 2022-01-25 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Period 1 (LY3410738 Alone) (Experimental): Single dose of LY3410738 administered orally.
  Interventions: Drug: LY3410738
- Part 1 Period 2 (LY3410738 + Itraconazole) (Experimental): Single dose of LY3410738 administered orally with multiple doses of itraconazole orally.
  Interventions: Drug: LY3410738; Drug: Itraconazole
- Part 2 Period 1 (LY3410738 Alone) (Experimental): Single dose of LY3410738 administered orally.
  Interventions: Drug: LY3410738
- Part 2 Period 2 (LY3410738 + Carbamazepine) (Experimental): Single dose of LY3410738 administered orally with multiple doses of carbamazepine orally.
  Interventions: Drug: LY3410738; Drug: Carbamazepine

INTERVENTIONS:
Drug: LY3410738 — Oral LY3410738
Drug: Itraconazole — Oral Itraconazole
  Arms: Part 1 Period 2 (LY3410738 + Itraconazole)
Drug: Carbamazepine — Oral Carbamazepine
  Arms: Part 2 Period 2 (LY3410738 + Carbamazepine)

SUMMARY:
The main purpose of this study is to learn about how itraconazole and carbamazepine affect the levels of LY3410738 in the blood stream of healthy participants. Participation could last up to 75 days.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential and males capable of fathering a child must use contraception
* Within body mass index (BMI) range 18.0 to 32.0 kilograms per square meter (kg/m²).
* Participants will be in good health, based on medical history, physical examination findings, vital signs, 12 lead electrocardiogram (ECG), or clinical laboratory tests, as determined by the Investigator (or designee).
* Able to comply with all study procedures, including the 15-night stay for those participating in part 1 or 25-night stay for those participating in part 2 at the Clinical Research Unit and follow-up phone call.

Exclusion Criteria:

* History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:

  1. Allergic disease
  2. Dermatological disease
  3. Renal disease
  4. Liver disease
  5. Pancreatitis
  6. Gastrointestinal disease
  7. Biliary disease
  8. Metabolic disease
  9. Hematological disease
  10. Pulmonary disease
  11. Neurological disease
  12. Cancer within the past 5 years
  13. Cardiovascular disease
* Participants with out-of-range, at-rest vital signs.
* Abnormal laboratory values determined to be clinically significant by the Investigator (or designee).
* Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination.
* Participation in any other investigational study drug trial involving administration of any investigational drug in the past 30 days or 5 half-lives, whichever was longer, prior to the first dose administration (Day 1).
* Use or intention to use any prescription or over-the-counter medications within 14 days or 5 half-lives (if known) prior to the first dose administration (Day 1) and through end of trial.
* History or presence of any illness or psychiatric condition, that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the participant at undue risk.
* Donation of blood from 56 days prior to Screening, plasma or platelets from 4 weeks prior to Screening.
* Receipt of blood products within 2 months prior to Check-in (Day -1).
* Significant history of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* For Part 1 only, Having impaired hearing or a history of hearing problems
* For Part 2 only, History of serious dermatological adverse reaction, such as toxic epidermal necrolysis, Stevens-Johnson syndrome, or DRESS
* For Part 2 only, Glaucoma or history of elevated intraocular pressure.
* For Part 2 only, Have answered 'yes' to either Question 4 or Question 3 on the 'Suicidal Ideation' portion of the Columbia Suicide Severity Rating Scale (C-SSRS) or have answered 'yes' to any of the suicide-related behaviors on the 'Suicidal Behavior' portion of the C-SSRS
* For Part 2 only, Have laboratory evidence of clinically significant anemia, leukopenia, thrombocytopenia, or hepatic dysfunction; or hyponatremia
* For Part 2 only, Genotyping test that is positive for either or both of the carbamazepine sensitivity conferring HLA alleles
* Creatinine clearance < 90 mL/minute calculated using the C-G equation at Screening or Check-in
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening, or evidence of such abuse as indicated by the laboratory assays for drugs of abuse (including cotinine and alcohol) conducted during Screening and/or at Check-in (Day- 1).
* Consumption of foods or beverages containing grapefruit/grapefruit juice or Seville oranges or their juice within 7 days prior to Check-in (Day -1) and through end of treatment (EOT) or early termination (ET)
* Have previously completed or withdrawn from this study or any other study investigating LY3410738, and have previously received LY3410738

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Assess the impact of multiple oral doses of itraconazole on single oral dose pharmacokinetics (PK) of LY3410738 by collecting/evaluating serum at protocol-specified time points: Maximum observed plasma concentration (Cmax) | Pre-dose up to 96 hours post-dose
  PK of LY3410738
Assess the impact of multiple oral doses of itraconazole on single oral dose PK of LY3410738 by collecting/evaluating serum at protocol-specified time points: Area under the concentration-time curve from Hour 0 to last measurable concentration (AUC0-t) | Pre-dose up to 96 hours post-dose
  PK of LY3410738
Assess the impact of multiple oral doses of itraconazole on single oral dose PK of LY3410738 by collecting/evaluating serum at protocol-specified time points: Area under the concentration-time curve extrapolated to infinity (AUC0-inf) | Pre-dose up to 96 hours post-dose
  PK of LY3410738
Assess the effect of multiple oral doses of carbamazepine on single oral dose PK of LY3410738 by collecting/evaluating serum at protocol-specified time points: Cmax | Pre-dose up to 96 hours post-dose
  PK of LY3410738
Assess the effect of multiple oral doses of carbamazepine on single oral dose PK of LY3410738 by collecting/evaluating serum at protocol-specified time points: AUC0-t | Pre-dose up to 96 hours post-dose
  PK of LY3410738
Assess the effect of multiple oral doses of carbamazepine on single oral dose PK of LY3410738 by collecting/evaluating serum at protocol-specified time points: AUC0-inf | Pre-dose up to 96 hours post-dose
  PK of LY3410738

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo, Study Director — Medical Monitor
Locations (1):
- LabCorp CRU, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No